CLINICAL TRIAL: NCT06654713
Title: Commercial or Open Source Closed Loop Impact on Pregnancy (COSCLIP) Study
Brief Title: Commercial or Open Source Closed Loop Impact on Pregnancy Study
Acronym: COSCLIP
Status: Recruiting | Type: Observational
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: 24-42036
Record Dates: First submitted 2024-10-15; First posted 2024-10-23 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Type 1 Diabetes; Pregnancy, High Risk; Insulin Dependent Diabetes; Pregnancy Related
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Commercial AID system: Pregnant individuals with type 1 diabetes (T1D) using commercially available automated insulin delivery (AID) systems for glycemic management in pregnancy
  Interventions: Other: Commercial AID system
- Open source AID system: Pregnant individuals with type 1 diabetes T1D) using open source automated insulin delivery (AID) systems (also known as do-it-yourself AID systems or hacked AID systems) for glycemic management in pregnancy
  Interventions: Other: Open source AID system

INTERVENTIONS:
Other: Commercial AID system — AID system that is commercially available and FDA approved for use
  Groups: Commercial AID system
Other: Open source AID system — AID system that uses unregulated open-source software to customize an insulin delivery algorithm to connect an insulin pump to a continuous glucose monitor
  Groups: Open source AID system

SUMMARY:
The goal of this observational study is to better understand what happens when pregnant people with type 1 diabetes (T1D) use automated insulin delivery (AID) systems. The main questions this study aims to answer are:

* What are the maternal and neonatal outcomes with AID system use in pregnancy?
* What are the glycemic outcomes with AID system use in pregnancy?
* What are the behavioral and emotional outcomes with AID system use in pregnancy?

Researchers will compare pregnant people who use commercial AID systems and pregnant people who use open source AID systems to see if outcomes are different with these different types of systems.

Participants will be asked to remotely share their AID system data with the research team; complete online surveys regarding behavioral and emotional health; and sign an authorization to release health information to allow the research team to access medical records.

ELIGIBILITY:
Inclusion criteria:

* Pregnant
* Diagnosis of type 1 diabetes (T1D) prior to pregnancy
* Active use of automated insulin delivery (AID) system

Exclusion criteria:

* Diagnosis of other forms of diabetes (gestational diabetes, type 2 diabetes, monogenic diabetes)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pregnant individuals with type 1 diabetes (T1D) using any form of automated insulin delivery (AID) system in pregnancy
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-03-13 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Large for gestational age (LGA) | At delivery
  Primary neonatal outcome. LGA defined as birth weight > 90th percentile for gestational age
Core score on Type 1 Diabetes Distress Assessment Scale (T1-DDAS) | From enrollment to 8 weeks postpartum
  Primary behavioral outcome. Score ranges from 1-5. Higher scores indicate higher degrees of diabetes distress.
Hypertensive disorders of pregnancy (HDP) | From enrollment to 8 weeks postpartum.
  Primary maternal outcome. As defined by the American College of Obstetricians and Gynecologists (ACOG).
Time in pregnancy-specific range (psTIR) | From enrollment to 8 weeks postpartum.
  Primary glycemic outcome. Defined as percent of time spent with sensor glucose in pregnancy range of 63-140 mg/dL.

SECONDARY OUTCOMES:
Incidence of cesarean delivery | At delivery
Incidence of neonatal hypoglycemia | From delivery to 28 days-of-life
Incidence of neonatal hyperbilirubinemia | From delivery to 28 days-of-life
Incidence of neonatal ICU admission | From delivery to 28 days-of-life
Incidence of major congenital malformations | From enrollment to delivery (up to 40 weeks of delivery)
Incidence of small for gestational age (SGA) | At delivery
  SGA defined as birth weight < 10th percentile for gestational age.
Incidence of pregnancy loss | From enrollment to delivery (up to 40 weeks of delivery)
Incidence of perinatal mortality | From delivery to 28 days-of-life
  Includes intrauterine fetal demise and neonatal demise
Incdience of diabetic ketoacidosis | From enrollment to 8 weeks postpartum
Incidence of maternal hypoglycemia | From enrollment to 8 weeks postpartum
Time above pregnancy-specific range (psTAR) | From enrollment to 8 weeks postpartum.
  Defined as percent of time spent with sensor glucose > 140 mg/dL.
Time spent below pregnancy-specific range (psTBR) | From enrollment to 8 weeks postpartum.
  Defined as percent of time spent with sensor glucose < 63 mg/dL.

CONTACTS AND LOCATIONS:
Overall Officials: Nasim Sobhani, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified IPD that underlie results in a publication
Time Frame: Beginning 6 months and ending 2 years after the publication of results